CLINICAL TRIAL: NCT06008691
Title: A Prospective, Observational Cohort Study to Evaluate the Clinical Impact of Novel Monoclonal Antibodies (MAB) in B-cell Non-Hodgkin Lymphoma (NHL) in Italian Clinical Practice
Brief Title: A Prospective, Observational Cohort Study on the Clinical Impact of Novel Monoclonal Antibodies in B-cell Non-Hodgkin Lymphoma in Italian Clinical Practice
Acronym: FIL_MAB
Status: Recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FIL_MAB
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma, B-cell
Keywords: Non-Hodgkin Lymphoma; B-cell; monoclonal antibodies; novel antibodies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Single Person

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- B-cell NHL patients treated with novel MAB in Italian real life (approved by EMA and AIFA).: B-cell NHL patients treated with novel MAB in Italian real life (approved by EMA since 2020 and prescribed according to the indications for use authorized for marketing in Italy).
  Patients first-line and relapsed or refractory who had received at least 1 dose of MAB.
  Different cohorts will be analyzed according to approved treatment indications, type of antibody employed and NHL hystotypes.
  Interventions: Drug: "novel" MAB (alone or in combination)

INTERVENTIONS:
Drug: "novel" MAB (alone or in combination) — "novel" MAB (alone or in combination) based on presence of an EMA clinical indication since 2020 and prescribed according to the indications for use authorized for marketing in Italy

SUMMARY:
This is a prospective, observational cohort study to evaluate the clinical impact of novel Monoclonal AntiBodies (MAB) in B-cell Non-Hodgkin Lymphoma (NHL) in Italian clinical practice.

DETAILED DESCRIPTION:
This is a large prospective, observational cohort study aimed at collecting clinical information on use, feasibility, short- and long-term efficacy and short- and long-term toxicity of novel MAB that have received approval from EMA since 2020 and are prescribed according to the indications for use authorized for marketing in Italy.

Patients entering the study will be subdivided into different cohorts based on approved treatment indications, type of antibody employed and histological subtype. Additional sub-cohorts will be defined if needed.

Final outputs will be based according to:

* Per indication analysis;
* Pooled analyses by type of antibody and subtype and other parameters;
* A general analysis of the whole cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of B-cell NHL and need of treatment (as per guideline indications), both first-line and relapsed or refractory.
* Patients aimed to be treated in indication with a "novel" MAB (alone or in combination) based on presence of an EMA clinical indication since 2020 and prescribed according to the indications for use authorized for marketing in Italy.
* Signed written informed consent.

Exclusion Criteria:

* Being involved in a prospective interventional trial outside indication.
* Patients treated outside approved indications:

  * 648-approved indication.
  * 5% AIFA support.
  * Compassionate use.
* Age less than 18 years.
* Inability to provide an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of B-cell NHL both first-line and relapsed or refractory aimed to be treated in indication with a "novel" MAB (alone or in combination) based on presence of an EMA clinical indication since 2020 and prescribed according to the indications for use authorized for marketing in Italy.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2038-10 (Estimated); Study Completion 2038-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | At least 5 years
  ORR will be defined according to Lugano 2014 criteria as the proportion of patients who have a partial response (PR) or complete response to therapy (CR+PR).
Complete Response rate (CRR) | At least 5 years
  CRR will be defined according to Lugano 2014 criteria and will include only patients who achieved a CR at the end of treatment program. The best overall response will be defined as the best response between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Progression free survival (PFS) | At least 5 years
  PFS is defined as the time between the date of enrollment and the first documentation of recurrence, progression or death from any cause; responding patients and patients who are lost to follow up will be censored at their last assessment date.
Overall survival (OS) | At least 5 years
  OS is defined as the time between the start of treatment until death from any cause; patients who are lost at follow up will be censored at their last assessment date.
Event free survival (EFS) | At least 5 years
  ESFS is defined as the time from start of treatment to disease progression, death, or discontinuation of treatment for any reason (e.g. toxicity, patient preference), or initiation of a new treatment without documented progression.
Time-to-next treatment (TTNT) | At least 5 years
  TTNT represents the interval from commencement of one treatment to initiation of the next line of therapy.
non-relapse mortality (NRM) | At least 5 years
  NRM is defined as death without recurrent or progressive disease after treatment.
Duration of response (DOR) | At least 5 years
  DOR is defined as the time from the first documentation of tumor response (CR/PR) to disease progression or death according to Lugano 2014 criteria.
Incidence of Early/Late Adverse Events | At least 5 years
  Toxicities will be recorded and classified according to the definitions of the latest version of the NCI CTCAE. Toxicity events will be determined by the incidence of severe, life-threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events (SAEs) commencing after the first induction dose or at any time during therapy. Early and toxic deaths and cause of any death. Special focus on second tumors, infections and autoimmune complications. Particularly:
  * Hematological and extra-hematological toxicities Grade > 2
  * Infusional adverse events, will be recorded any Grade
  * Toxicities of specific interest on second tumors, infections and autoimmune complications will be recorded any Grade
  * Early and toxic deaths and cause of any death.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ladetto, Prof., Principal Investigator — AO SS Antonio e Biagio e Cesare Arrigo, Alessandria
Locations (61):
- Italy (61):
  - Istituto Oncologico del Mediterraneo SPA - Oncologico, Viagrande, Catania
  - Ospedale SS. Cosma e Damiano - Ospedale San Jacopo - SOS Oncoematologia ed ematologia clinica, Pescia, Pistoia
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia, Alessandria
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - IRCCS Centro di Riferimento Oncologico di Aviano - Divisione di Oncologia e dei Tumori immuto-correlati, Aviano
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia, Bari
  - Ospedale "Monsignor Raffaele Dimiccoli" - Ematologia, Barletta
  - Azienda Ospedaliera Papa Giovanni XXIII - Ematologia, Bergamo
  - Nuovo Ospedale degli Infermi - SSD Ematologia, Biella
  - Policlinico S. Orsola-Malpighi - Istituto di Ematologia "Seragnoli", Bologna
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Businco - SC Ematologia e CTMO, Cagliari
  - Fondazione del Piemonte per l'Oncologia - IRCCS - Ematologia, Candiolo
  - Osp. civile di Carrara - Oncologia Medica, Carrara
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - Arnas Nuovo Ospedale Garibaldi Nesima - U.O.C. Ematologia, Catania
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco - UOC di Emtologia, Catania
  - Ospedale di Civitanova Marche - UOSD EMATOLOGIA AREA VASTA 3 MACERATA, Civitanova Marche
  - ASST Cremona - Ematologia e CRTO, Cremona
  - A.O. S. Croce e Carle - S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Presidio Ospedaliero F. Spaziani - UOC Ematologia, Frosinone
  - Ospedale Versilia USL NORDOVEST Toscana - UOS Ematologia, Lido di Camaiore
  - Ospedale di Livorno - Ematologia, Livorno
  - Ospedale Apuane - Oncoematologia, Massa
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - ASST Santi Paolo e Carlo - Onco - Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - Istituto Scientifico San Raffaele - Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori - Ematologia, Monza
  - AOU Federico II - Ematologia, Napoli
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto - U.O. Ematologia, Piacenza
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - Ospedale S.Stefano SOS Oncoematologia, Prato
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - IRCCS-Centro di Riferimento Oncologico - UO di ematologia e Trapianto Cellule Staminali, Rionero in Vulture
  - AO Sant' Andrea - Ematologia, Roma
  - Policlinico Umberto I - Università "La Sapienza" - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Roma
  - Policlinico Universitario Campus Bio-Medico - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano
  - AOU di Sassari - Ematologia, Sassari
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - AOU Senese - U.O.C. Ematologia, Siena
  - Ospedale "G. Mazzini" - UOS Ematologia, Teramo
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O.U. Città della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - Ospedale Ca' Foncello - S.C di Ematologia, Treviso
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ematologica, Udine
  - AOU Integrata di Verona - U.O. Ematologia, Verona
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza